CLINICAL TRIAL: NCT01347515
Title: Bioavailability and Bioactivity of Olive Oils Enriched With Their Own Phenolic Compounds in a Dose-response Study (VOHF1)
Brief Title: Bioactivity of Olive Oils Enriched With Their Own Phenolic Compounds (VOHF1)
Acronym: VOHF1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Rovira i Virgili (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government); Universitat de Lleida (Other); Fundacion IMIM (Other)
Responsible Party: Rosa SOLÀ, URoviraiVirgili
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: URoviraiVirgili
Record Dates: First submitted 2011-04-26; First posted 2011-05-04 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-04

CONDITIONS: Polyphenol Absorption in Healthy People
Keywords: Phenol-enriched olive oil; bioavailability; bioactivity
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FOO250 (Placebo Comparator): FOO250 ppm, the standard virgin olive oil
  Interventions: Other: olive oil
- FOO500 (Active Comparator): Olive oil enriched with its own broad-spectrum phenolic compounds; FOO500 ppm
  Interventions: Other: olive oil
- FOO750 (Active Comparator): Olive oil enriched with its own broad-spectra phenolic compounds; FOO750 ppm
  Interventions: Other: olive oil

INTERVENTIONS:
Other: olive oil — Each volunteer will be given, in random order, a single dose of 30 ml on a base of 80 g bread, of the following functional olive oils (FOO): FOO750 ppm, FOO500 ppm, which are enriched with two different amounts of broad-spectrum phenolic compounds from the virgin FOO250 ppm; all prepared at the Universitat de Lleida.
  Post-ingestion the volunteers will rest for 8h in a comfortable warm room. During the run-in period of 2 weeks prior the first postprandial study and 1 week between each FOO treatment period, all subjects will undergo a 2-day pre-treatment wash-out period of a phenol-free diet (saturated fatty acids in the diet will be 10-13% of energy in an isocaloric diet). Volunteers will avoid non-essential physical activity during the 3 days prior to the treatment day.
  Other Names: Functional olive oil

SUMMARY:
Hypothesis: A functional olive oil tailored to provide the best relationship between phenolic compounds (amount and type) phenolic bioavailability and bioactivity (antioxidant and anti-endothelial dysfunction) will be a useful tool for increasing not only circulating HDL cholesterol concentration, but also the functionality (antioxidant, anti-inflammatory, and reverse cholesterol transport capacity) of human HDL in vivo.

DETAILED DESCRIPTION:
The first step is to determine, in healthy human subjects in postprandial condition, the best relationship between phenolic compounds (amount and type) / bioavailability and bioactivity (antioxidant, anti-inflammatory and anti-endothelial dysfunction) using olive oils enriched with its own broad-spectrum phenolic compounds.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers aged 20 to 70 years

Exclusion Criteria:

1. LDL cholesterol levels above 189 mg/dL
2. Triglycerides ≥350 mg/dL (the upper limit for correctly determining LDL-c by the Friedewald formula)
3. Physical examination and routine biochemical laboratory determinations will be carried out to exclude co-morbidities
4. Intake of antioxidant supplement or acetylsalicylic acid or any other drug with known antioxidative properties
5. Chronic alcoholism
6. Body mass index (BMI)≥30 kg/m2
7. Statin treatment prior to initiating the trial; stopped at least 2 months before starting the study
8. Antihypertensive treatment prior to initiating the trial; stopped at least 2 months before starting the study
9. Diabetes mellitus (fasting blood glucose > 126 mg/dL; measurements repeated for confirmation)
10. Renal disease (plasma creatinine levels > 1.4 mg/dL for women and > 1.5 mg/dL for men
11. Acute infectious diseases, malignancies, severe liver insufficiency, chronic respiratory insufficiency or associated endocrine diseases
12. Other conditions with special nutritional requirements
13. Having participated in a clinical trial in the last 3 months, or currently participating in a clinical trial
14. Inability to continue in the study
15. History of gastrointestinal disease that can impair the absorption of nutrients
16. Depression syndrome or self-injuring ideation
17. High plasma C-reactive protein and ESR concentrations
18. Immunization in the last 2 months
19. Anemia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Changes in the dose-response study with olive oils (FOO250, FOO500 and FOO750) enriched with broad-spectrum phenolic compounds | Changes from baseline (pre-ingestion) in Bioavailability of phenolic compounds at 8h after olive oil intake
  Bioavailability of phenolic compounds from olive oils in plasma and urine until 8h post olive oil-intake.

SECONDARY OUTCOMES:
Changes of bioactivity with olive oild (FOO250, FOO500 and FOO750)enriched with broad-spectrum phenolic compounds | Changes form baseline (pre-ingestion) in endothelial function of phenolic compounds at 6h after olive oil
  Endothelial function will be measured through the assessment of ischemic reactive hyperemia (IRH), at baseline and at 2h, 4 h and 6 after olive oil intake
Changes in bioactivity of FOO250, FOO500 and FOO750 | Changes form baseline (pre-ingestion) at 6h or 8h after oral olive oil intake in bioactivity
  Biomarkers of cardiovascular disease: Oxidative; Lipid profile; Insulin resistance; Inflammation biomarkers; Endothelial dysfunction; Anti-thrombotic activity; Identification and quantification in human plasma and in urine of phenol metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, MD, PhD, Principal Investigator — Universitat Rovira i Virgili, Spain
Locations (1):
- Hospital Universitari Sant Joan, Universitat Rovira i Virgili, Reus, Tarragona, Spain